CLINICAL TRIAL: NCT00203931
Title: A Randomized Phase II Trial Comparing Cetuximab With Concurrent Pemetrexed/Cetuximab Therapy for Non-Small Cell Lung Cancer Refractory to Primary Treatment
Brief Title: Trial Comparing Cetuximab With Pemetrexed/Cetuximab Therapy for Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual and evidence from other studies showing benefit of early initiation of pemetrexed after first-line therapy
Sponsor: University of Chicago (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13722A
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Results first posted 2014-03-31 (Estimated); Last update posted 2014-03-31 (Estimated); Status verified 2014-02

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cetuximab; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cetuximab (Active Comparator): Cetuximab initial dosage of 400 mg/m2 over 120 minutes, followed by weekly infusions at 250 mg/m2 over 60 minutes.
  Interventions: Drug: Cetuximab
- Cetuximab and Pemetrexed (Experimental): Cetuximab initial dosage of 400 mg/m2 over 120 minutes, followed by weekly infusions at 250 mg/m2 over 60 minutes. Starting on day 15 and then subsequently on day 1 of each 21 day cycle, Pemetrexed 500 mg/m2.
  Interventions: Drug: Cetuximab; Drug: Pemetrexed

INTERVENTIONS:
Drug: Cetuximab
  Other Names: ERBITUX
Drug: Pemetrexed
  Other Names: ALIMTA
  Arms: Cetuximab and Pemetrexed

SUMMARY:
The purpose of the study is to determine in patients with Non Small Cell Lung Cancer refractory to previous chemotherapy whether concomitant treatment with cetuximab and pemetrexed improves progression-free survival compared with cetuximab monotherapy.

DETAILED DESCRIPTION:
While EGFR inhibitors have demonstrated activity against NSCLC [their integration into first-line therapy in combination with standard agents has yielded disappointing results]. There are many potential reasons for the disappointing results in these first-line studies [ A single-arm Phase I trial of cetuximab in combination with docetaxel suggested better efficacy in second-line therapy for NSCLC than docetaxel alone but this comes at the expense of some increased toxicity]. Preliminary data indicate that cetuximab has single agent activity in this setting. The confidence intervals for this activity overlap the median time to progression of the current second-line cytotoxic therapy options compared in the Hanna study [A clinically relevant question is- does concurrent cetuximab and pemetrexed significantly improve upon outcomes of cetuximab monotherapy followed by pemetrexed monotherapy?].

Many patients who receive EGFR inhibitors develop an acneiform rash and the severity of the rash is associated with good outcomes from treatment. Several of these studies have demonstrated no correlation between the intensity or percentage of tumor cells staining for EFUR expression and response to therapy. However, a Phase II study, at the University of Colorado, of cetuximab added to standard first-line treatment of NSCLC revealed 6/10 responders developed the rash within 2 weeks of initiating treatment (Personal Communication, Dugan, et al. BMS). Therefore, early development of rash may be a clinically useful marker of subsequent response and novel approaches to the identification of biological markers for this phenotype prior to initiation of therapy may be helpful in subsequent determination of which patients will most likely benefit from EGFR inhibitor therapy.

To address these issues we propose a phase I randomized study of concurrent pemetrexed/cetuximab compared to sequential cetuximab/pemetrexed therapy for the second-line treatment of advanced NSCLC. Patients will be randomized at study entry. Regarding prospective analysis of the rapid-rash forming phenotype, all patients will receive 2 weeks of initial treatment with cetuximab and undergo formal rash evaluation, serum and skin collection. According to the initial randomization, half of the study subjects will continue with cetuximab monotherapy while the remainder will receive concurrent cetuximab and pemetrexed. The primary study endpoint of freedom from progression and secondary endpoint of objective response rate will be based on the comparison of patients in (he concurrent therapy group with patients treated with cetuximab monotherapy with Day-14 (first receipt of cetuximab) as the reference treatment start date. Overall survival will be analyzed as a secondary endpoint to assess the efficacy of concomitant treatment with cetuximab and pemetrexed compared to sequential treatment with cetuximab followed by pemetrexed upon disease progression. As patients in both treatment arms receive cetuximab, correlative studies will be performed on all enrolled patients. For serum proteomic studies designed to identify a serum polypeptide signature associated with response to cetuximab-based therapy, serum samples shall be collected at enrollment, and just prior to receiving the third dose of cetuximab therapy. To provide the opportunity to perform retrospective pharmacogenomic studies, whole blood DNA will be collected from each patient at enrollment and subsequently analyzed for candidate gene polymorphisms once outcome data is available. Finally, an alternative approach to identification of markers for responsiveness to EGFR inhibition already in progress at the University of Chicago entails collection of skin biopsies before and after treatment with an EGFR inhibitor.

As in ongoing collaborations with the University of Chicago Section of Dermatology, patients in this proposed study will undergo skin biopsies at enrollment and after 2 weeks of cetuximab therapy. The investigators will extract mRNA from the fresh frozen skin specimens and perform microarray studies to test the utility of mRNA expression patterns associated with rash and responsiveness to EOFR inhibitors in currently ongoing investigations at the University of Chicago. Therefore we expect this study: 1) to identify any significant improvement of concurrent cetuximab/pemetrexed therapy for second-line treatment of NSCLC over sequential monotherapy, 2) through timely minimally invasive collection of serum and exposed skin, to provide the opportunity to test previously identified biomarkers for individual responsiveness to cetuximab therapy, and 3) to confirm prospectively whether early development of rash on cetuximab treatment predicts responsiveness to either concurrent or sequential therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of locally advanced or metastatic (Stage III or IV at entry) non-small cell lung cancer (NSCLC) that is not amenable to curative therapy.
* ECOG performance status 0-2
* Patients must have been previously treated with one platinum-containing or taxane-containing chemotherapy regimen for locally advanced or metastatic disease. Patients are also eligible if they have received one platinum-based chemotherapy regimen as neoadjuvant or adjuvant chemotherapy, but must have received an additional chemotherapy regimen upon recurrence.
* No more than two prior systemic anti-cancer therapies will be allowed.
* Prior radiation therapy is allowed to <25% of the bone marrow. Prior radiation to the whole pelvis is not allowed, Prior radiotherapy must be completed at least 2 weeks before study enrollment, and the patient must have recovered from the acute toxic effects of the treatment prior to study enrollment.
* Patients must have signed an approved informed consent.
* Male and female patients with reproductive potential must use an approved contraceptive method if appropriate (eg, intrauterine device, birth control pills, or barrier device) during and for 3 months after the study. Female patients must either not be of child bearing potential or have a negative pregnancy test within 7 days of treatment. Patients are considered not of child bearing potential if they are surgically sterile (they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are postmenopausal.
* Age>18
* Measurable disease in accord with RECIST criteria
* Bone marrow Function: absolute neutrophil count (ANC)>/=1,500/ul, platelets >/=l00,000, hemoglobin> 9g/dL
* Renal function: creatinine clearance (calculated by Cockcroft and Gault method) >/= 45mL/min
* Hepatic function: bilirubin </=1.5 x ULN; ALT/AST ,/= 2.5 x ULN; Albumin >/=2.5 g/dL

Exclusion Criteria:

* Prior treatment with pemetrexed
* Prior therapy that targets the EGF pathway.
* Active or uncontrolled infection.
* Significant history of uncontrolled cardiac disease; i.e., uncontrolled hypertension, unstable angina, and congestive heart failure.
* Pleural or pericardial effusions that cannot be completely evacuated prior to pemetrexed therapy.
* Acute hepatitis or known HIV.
* Prior severe infusion reaction to a monoclonal antibody.
* Any concurrent chemotherapy not indicated in the study protocol or any other investigational agent(s).
* Pregnancy or Breast-feeding.
* Second primary malignancy that is clinically detectable at the time of consideration for study enrollment.
* Inability to interrupt aspirin, or other nonsteroidal anti-inflammatory agents for a 5-day period.
* Inability or unwillingness to take folic acid or vitamin B12 supplementation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2005-03; Primary Completion 2008-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Maitland, M.D., Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Maitland ML, Levine MR, Lacouture ME, Wroblewski KE, Chung CH, Gordon IO, Szeto L, Ratko G, Soltani K, Kozloff MF, Hoffman PC, Salgia R, Carbone DP, Karrison TG, Vokes EE. Evaluation of a novel rash scale and a serum proteomic predictor in a randomized phase II trial of sequential or concurrent cetuximab and pemetrexed in previously treated non-small cell lung cancer. BMC Cancer. 2014 Jan 4;14:5. doi: 10.1186/1471-2407-14-5. PMID 24386952

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cetuximab | Cetuximab and Pemetrexed
Started | 27 | 28
Completed | 20 (These are the evaluable patients who received at least 3 doses of cetuximab.) | 23 (These are the evaluable patients who received at least 3 doses of cetuximab.)
Not Completed | 7 | 5

BASELINE CHARACTERISTICS:
Population: Includes evaluable patients (those that received at least 3 doses of cetuximab)
Groups:
- Total: Total of all reporting groups
Arm/Group | Cetuximab | Cetuximab and Pemetrexed | Total
Number analyzed (Participants) | 20 | 23 | 43
Age, Continuous [Median (Full Range); unit: years] | 62 [36 to 76] | 55 [45 to 75] | 58 [36 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 16
  Male | 14 | 13 | 27
Region of Enrollment [Number; unit: participants]
  United States | 20 | 23 | 43

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression-free survival will be defined as the time from the start of treatment until progression (documented according to Response Evaluation Criteria in Solid Tumors [RECIST] criteria and defined as at least a 20% increase in the sum of the longest diameter of target lesions) or death from any cause, whichever comes first.
Time Frame: Up to 5 years
Population: Includes evaluable patients (those that received at least 3 doses of cetuximab)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab | Cetuximab and Pemetrexed
Number analyzed (Participants) | 20 | 23
months | 1.6 [0.9 to 1.9] | 2.3 [1.6 to 3.1]
Statistical Analysis 1: Comparison: Cetuximab vs Cetuximab and Pemetrexed; Test type: Superiority or Other; p = 0.11, Log Rank

2. Secondary Outcome: Progression-free Survival Based on Rash Development
Description: Progression-free survival in this landmark analysis looking at the utility of early rash in predicting progression-free survival will be defined as the time from day 22 of study therapy until progression (documented according to Response Evaluation Criteria in Solid Tumors [RECIST] criteria and defined as at least a 20% increase in the sum of the longest diameter of target lesions) or death from any cause, whichever comes first. Patients last known to be alive and progression-free were censored at the date of the last scan without evidence of progression.
Time Frame: up to 5 years
Population: Includes evaluable patients (those that received at least 3 doses of cetuximab), but the total number analyzed is not 43 because 2 patients died or progressed prior to day 22 of cetuximab therapy and thus were excluded from this analysis.
Measure: Median (Standard Error); unit: months
Groups:
- Early Rash: Presence of rash (grade 1 or higher) by day 21 of cetuximab therapy
- No Early Rash: Absence of rash (grade 1 or higher) by day 21 of cetuximab therapy
Arm/Group | Early Rash | No Early Rash
Number analyzed (Participants) | 37 | 4
months | 0.9 (0.1) [0.9 to 2.0] | 0.9 (0.5) [lower limit 0.03]
Statistical Analysis 1: Comparison: Early Rash vs No Early Rash; Test type: Superiority or Other; p = 0.91, Wilcoxon-Gehan test

3. Secondary Outcome: Objective Response Rate
Description: Objective response (complete response [CR] + partial response [PR]) will be evaluated using RECIST criteria. CR is the disappearance of all target lesions. PR requires at least a 30% decrease in the sum of the longest diameter of target lesions.
Time Frame: up to 2 years
Population: Includes evaluable patients (those that received at least 3 doses of cetuximab).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab | Cetuximab and Pemetrexed
Number analyzed (Participants) | 20 | 23
percentage of participants | 0 [0 to 16.8] | 13.0 [2.8 to 33.6]
Statistical Analysis 1: Comparison: Cetuximab vs Cetuximab and Pemetrexed; Test type: Superiority or Other; p = 0.24, Fisher Exact

4. Secondary Outcome: Overall Survival
Description: Overall survival will be defined as the time from the start of treatment until death from any cause.
Time Frame: Up to 5 years
Population: Includes evaluable patients (those that received at least 3 doses of cetuximab)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab | Cetuximab and Pemetrexed
Number analyzed (Participants) | 20 | 23
months | 3.5 [2.8 to 11.7] | 10.3 [7.5 to 16.8]
Statistical Analysis 1: Comparison: Cetuximab vs Cetuximab and Pemetrexed; Test type: Superiority or Other; p = 0.046, Wilcoxon-Gehan test

5. Secondary Outcome: Progression-free Survival Based on Serum Biomarker Status
Description: Progression-free survival in this analysis looking at the association between a serum proteomic biomarker and progression-free survival will be defined as the time from the start of treatment until progression (documented according to Response Evaluation Criteria in Solid Tumors [RECIST] criteria and defined as at least a 20% increase in the sum of the longest diameter of target lesions) or death from any cause, whichever comes first.
Time Frame: up to 5 years
Population: Includes evaluable patients (those that received at least 3 doses of cetuximab), but the total number analyzed is not 43 because 10 patients did not have a pre-treatment/baseline serum marker classification and thus were excluded from this analysis.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Poor Prognosis; Good Prognosis: VeriStrat assigned classification based on mass spectrometry-based assay of serum samples collect at baseline. Details of how this was done is provided in "Mass spectrometry to classify non-small-cell lung cancer patients for clinical outcome after treatment with epidermal growth factor receptor tyrosine kinase inhibitors: a multicohort cross-institutional study." by Taguchi et al. in J Natl Cancer Inst 2007 99(11): 838-46.
Arm/Group | Poor Prognosis | Good Prognosis
Number analyzed (Participants) | 12 | 21
months | 1.57 [0.7 to 1.9] | 1.64 [1.6 to 3.3]
Statistical Analysis 1: Comparison: Poor Prognosis vs Good Prognosis; Test type: Superiority or Other; p = 0.029, Log Rank

ADVERSE EVENTS:
Time Frame: up to 5 years
Description: Serious adverse events of any grade are reported. For all other adverse events, only those grade 3 or higher were collected during the study. Adverse events are reported for the evaluable patients who received at least 3 doses of Cetuximab
Arm/Group | Cetuximab | Cetuximab and Pemetrexed
Serious Adverse Events (participants affected / at risk) | 11/20 | 7/23
Other Adverse Events (participants affected / at risk) | 15/20 | 17/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab (N=20) | Cetuximab and Pemetrexed (N=23)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Cataract (Eye disorders) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Pain (General disorders) | 2 | 1
Fever (General disorders) | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Superior vena cava syndrome (Vascular disorders) | 0 | 1
Vasovagal reaction (Nervous system disorders) | 1 | 0
Confusion (Psychiatric disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Infection (Infections and infestations) | 2 | 2
Neutrophil count decreased (Investigations) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 1 | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab (N=20) | Cetuximab and Pemetrexed (N=23)
Fatigue (General disorders) | 5 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 11 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes